CLINICAL TRIAL: NCT02106910
Title: Non-Endoscopic Surveillance for Barrett's Esophagus Following Ablative Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Cambridge (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-2618; 1K24DK100548-01 (NIH)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-07

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Radiofrequency Ablation
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Participants with Barrett's and No History of Ablation (Experimental): Participants with a diagnosis of BE, presenting for routine care endoscopy for surveillance or treatment of their BE.
  Interventions: Device: Cytosponge
- Participants with Barrett's and a History of Ablation (Experimental): Participants with Barrett's Esophagus (BE) with low grade dysplasia (LGD) or high grade dysplasia (HGD) and achieved complete eradication of BE via radiofrequency ablation (RFA).
  Interventions: Device: Cytosponge

INTERVENTIONS:
Device: Cytosponge — The Cytosponge is a simple, non-endoscopic device developed for endoscopic screening of subjects at risk for Barrett's esophagus (BE) by investigators at the University of Cambridge in the U.K. The Cytosponge is an ingestible gelatin capsule enclosing a compressed spherical polyurethane mesh sponge of 3 cm diameter, the center of which is attached to a string (Astralen, braided synthetic non-absorbable suture) (Figure 1). The capsule and string are swallowed with water. The string is held at the mouth without tension by means of a 7 cm cardboard tab attached to the string, and esophageal peristalsis and gravity move the capsule into the stomach. After 5 to 7 minutes (during which the gelatin capsule dissolves and the sponge is liberated), the sponge is withdrawn by gentle traction on the string and as it does so, collects cells from the lining of the esophagus. The sponge is placed in fixative for 48 hours, then the cells are pelleted, and processed into paraffin blocks

SUMMARY:
Subjects presenting to University of North Carolina at Chapel Hill (UNC) Hospitals for routine endoscopic surveillance examinations for current Barrett's Esophagus (BE) or after successful radiofrequency ablation (RFA) of dysplastic Barrett's Esophagus (BE) will be offered enrollment in the study. After informed consent, and the same day as the endoscopic procedure, the subject will undergo administration of the Cytosponge assay. The patient will then undergo routine endoscopic surveillance, using a standard Seattle biopsy surveillance protocol. The Cytosponge will be placed in fixative and shipped to the Fitzgerald laboratory at the University of Cambridge for processing according to their established protocols. Tissue biopsies will undergo standard processing and Hematoxylin and Eosin (H&E) staining, with assessment by expert gastrointestinal pathologists at UNC. The primary outcome variables will be sensitivity and specificity of the novel assay, compared against the gold standard of the presence of recurrent BE as detected by upper endoscopy with biopsies. Secondary outcomes include acceptability of the nonendoscopic assay to the patient (assessed by a standardized tool, the Impact of Events Scale, as well as a visual analogue scale), and likelihood of assay positivity as a function of amount of residual disease (as measured by Prague criteria).

DETAILED DESCRIPTION:
Esophageal Adenocarcinoma is a Lethal Cancer with a Rapidly Increasing Incidence. Barrett's Esophagus (BE) is the Strongest Risk Factor for Esophageal Adenocarcinoma. Endoscopic Ablation Induces Reversion of Barrett's Esophagus, and Decreases Progression of Disease. Unfortunately, data demonstrate a risk of recurrence of BE following successful eradication. Recent data published by the candidate and colleagues from the Ablation of Intestinal Metaplasia Containing Dysplasia (AIM Dysplasia) study demonstrate that approximately 25% of subjects who experience successful eradication of dysplastic BE will develop recurrent BE.

Therefore, following successful endoscopic ablation, patients receive ongoing endoscopic surveillance. More recently, a simple, non-endoscopic device, termed the Cytosponge, has been developed for endoscopic screening of subjects at risk for BE. Cytosponge demonstrated a sensitivity of 90% and a specificity of 94% for the detection of BE.

We expect these investigations to lead to a less costly, highly accurate, less invasive and more preferred screening paradigm for the large number of subjects who have undergone endoscopic ablative therapy.

The Cytosponge is a simple, non-endoscopic device developed for endoscopic screening of subjects at risk for Barrett's esophagus (BE) by investigators at the University of Cambridge in the U.K. The Cytosponge is an ingestible capsule enclosing a compressed spherical mesh sponge of 3 cm diameter, the center of which is attached to a string. The capsule and string are swallowed with water. The string is held at the mouth without tension by means of a cardboard tab attached to the string, and esophageal peristalsis and gravity move the capsule into the stomach. After 5 minutes (during which the capsule dissolves and the sponge is liberated), the sponge is withdrawn by gentle traction on the string and as it does so, collects cells from the lining of the esophagus. The sponge is placed in fixative, then the cells are pelleted, and processed into paraffin blocks. The pellets are immunostained with trefoil factor 3, which is interpreted simply as either positive or negative by the presence of any staining.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18-80 years,
2. Meets the following:

   2.1. Previous diagnosis of Barrett's Esophagus (BE) with dysplastic low grade dysplasia (LGD) or high grade dysplasia (HGD), as evidenced by both classical endoscopic appearance of salmon-colored mucosa in the tubular esophagus, as well as endoscopic biopsies from the involved areas demonstrating columnar metaplasia with goblet cells. The diagnosis of dysplasia must have been confirmed by a second expert pathologist. Previous endoscopic mucosal resection (EMR) of focal nodular high grade dysplasia (HGD) or superficial intramucosal cancer (IMC) is allowable, as long as the EMR specimen shows complete resection of any IMC with clear margins, and biopsies following ablation confirm excision of the lesion, AND 2.1.1. A history of complete eradication of both dysplasia and intestinal metaplasia by radiofrequency ablation. Complete eradication is defined as a normal endoscopic appearance of the tubular esophagus, and histologic confirmation by biopsies in 4 quadrants every cm from throughout the length of the previous BE (post-RFA cohort).OR 2.2. Current diagnosis of BE, presenting for routine care endoscopy (BE cohort).
3. Good general health, with no severely debilitating diseases, active malignancy, or condition that would interfere with study participation.

Exclusion Criteria:

1. Current use of blood thinners such as coumadin, warfarin, clopidogrel, heparin and/or low molecular weight heparin (requires discontinuation of medication 5 days prior to and 7 days after esophagogastroduodenoscopy (EGD) and Cytosponge administration, aspirin use is OK).
2. Known bleeding disorder
3. For the post-RFA cohort, prior ablative therapy of the esophagus other than radiofrequency ablation (RFA), including photodynamic therapy (PDT), more than one session of spray cryotherapy, and any other ablation therapies is exclusionary. However, prior endoscopic mucosal resection (EMR) is acceptable and up to two prior treatments of thermal/coagulation therapy (other than RFA) for focal residual disease following otherwise successful RFA therapy is acceptable.
4. History of esophageal stricture precluding passage of the endoscope or sponge,
5. Pregnancy, or planned pregnancy during the course of the study,
6. Any history of esophageal varices, liver impairment of moderate or worse severity (Child's- Pugh class B & C) or evidence of varices noted on any past endoscopy,
7. Any history of esophageal surgery, except for uncomplicated fundoplication, and,
8. History of coagulopathy, with international normalized ratio (INR) >1.3 and/or platelet count of <75,000.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Barrett's and no History of Ablation: Participants presenting with Barrett's Esophagus (BE) for routine endoscopic examinations with no history of ablation.
  Cytosponge Cell Collection Device is indicated for use in the collection and retrieval of surface cells in the esophagus.
- Participants With Barrett's After Ablation: Participants presenting with Barrett's Esophagus (BE) for routine endoscopic examinations after history of at least one session of Endoscopic Eradiation Therapy (EET).
  Cytosponge Cell Collection Device is indicated for use in the collection and retrieval of surface cells in the esophagus.
Period: Overall Study
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
Started | 49 | 89
Completed | 48 | 88
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation | Total
Number analyzed (Participants) | 49 | 89 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (10.6) | 66.3 (8.8) | 65.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 36 | 71 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 49 | 88 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 89 | 138

OUTCOME MEASURES:

1. Primary Outcome: Cytosponge Acceptability by Number of Participants
Description: Acceptability will be measured the Impact of Events Scale (IES). This scale was developed to assess the distress associated with a specific life event. Respondents are asked to answer questions to indicate the amount of stress from the event. Scores are calculated with the following scale, (Not at all =0, Rarely =1, Sometimes =3, Often =5). Assessment yields a cumulative score that are calculated from each response, with a total final score ranging from (0-75). High scores represent high test induced distress and lower values represent low distress.
Time Frame: 7 days after Baseline
Population: Data unavailable for 2 participants who did not complete assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Barrett's After Ablation: Participants presenting with Barrett's Esophagus (BE) for routine endoscopic examinations after history of at least one session of Endoscopic Eradiation Therapy (EET).
  Cytosponge Cell Collection Device is indicated for use in the collection and retrieval of surface cells in the esophagus.
  Period Title: Overall Study
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
Number analyzed (Participants) | 48 | 88
Participants
  No meaningful impact (Scores 0-8) | 46 | 81
  Impact Event (Scores 9-25) | 2 | 6
  Powerful Impact Event (Scores 26-43) | 0 | 1
  Severe Impact Event (Scores 44-75) | 0 | 0

2. Primary Outcome: Mean Post Procedure Pain on the Visual Analog Scale
Description: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 100-mm line that represents a continuum between "no pain" and "worst pain." Higher scores are representative of worse pain.
Time Frame: Immediately after Cytosponge removal
Population: Data unavailable for 2 participants who did not complete assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
Number analyzed (Participants) | 48 | 88
units on a scale | 19.1 (17.7) | 17.0 (17.5)

3. Primary Outcome: Willingness to Repeat Cytosponge by Number of Participants
Description: Participants were asked if they would be willing to repeat the Cytosponge, yes/no.
Time Frame: 7 days after Baseline
Population: Data unavailable for 3 participants who did not complete assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
Number analyzed (Participants) | 47 | 88
Participants
  Yes | 44 | 86
  No | 3 | 2

4. Primary Outcome: Mean Procedure Preference Rating
Description: Participants were asked to rate both procedures (Cytosponge and esophagogastroduodenoscopy (EGD)) to indicate which procedure they preferred on a scale from 0-10. Higher scores represent greater preference.
Time Frame: 7 days after Baseline
Population: Data unavailable for 2 participants who did not complete assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
Number analyzed (Participants) | 48 | 88
Units on a scale
  Cytosponge Rating, On scale of 1-10 | 7.8 (2.3) | 7.9 (2.0)
  EGD Rating, On scale of 1-10 | 9.2 (1.4) | 9.1 (1.5)

5. Secondary Outcome: Cytosponge™ Operating Characteristics
Description: The operating characteristics of the Cytosponge™ technique compared against a gold standard of upper endoscopy with biopsies for endoscopic surveillance was evaluated for sensitivity and specificity in the detection of BE in subjects with current (BE) or history of successful radiofrequency ablation for dysplastic BE. A true positive was considered when both the endoscopic biopsy and the Cytosponge detected the goblet cells characteristic of BE. A false positive was considered when the Cytosponge demonstrated these cells while the biopsies did not. A true negative occurred when neither the biopsies nor the Cytosponge showed goblet cells. A false negative was considered when the biopsies did demonstrate goblet cells while the Cytosponge did not. True Positives (TP) and False Negatives calculate sensitivity: (TP)/(TP + FN); True Negatives (TN) and False Positives (FP) are used to calculate specificity: (TN)/(TN + FP).
Time Frame: Baseline
Population: Data unavailable for 2 participants who did not complete assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
Number analyzed (Participants) | 48 | 88
percentage of participants
  Specificity to detect BE | 92.00 | 85.00
  Sensitivity to detect BE | 80.00 | 74.00
  Assay Accuracy | NA — Analysis not available. | 84.00

ADVERSE EVENTS:
Time Frame: From Baseline until approximately 30 days after completion of biomarker panel, an overall approximate total of 45 days.
Description: Per study protocol section 7.2, only those events that are potentially related to participation in this research study must be reported.
Arm/Group | Participants With Barrett's and no History of Ablation | Participants With Barrett's After Ablation
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/89
Other Adverse Events (participants affected / at risk) | 7/49 | 14/89
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Barrett's and no History of Ablation (N=49) | Participants With Barrett's After Ablation (N=89)
Sore Throat (Gastrointestinal disorders) | 7 (7) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT02106910/Prot_SAP_000.pdf